CLINICAL TRIAL: NCT03835299
Title: Addressing Fear and Risk of Vasovagal Reactions Among High School Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: New York Blood Center (Other)
Responsible Party: Principal Investigator, Christopher R. France, Ph.D., Distinguished Professor of Psychology, Ohio University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NYBC 1243761
Record Dates: First submitted 2019-02-07; First posted 2019-02-08 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Blood Donors
Keywords: blood donor, fear, vasovagal reaction
MeSH Terms: conditions — Syncope, Vasovagal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators are masked because the participants are randomized and the intervention is delivered by a computer tablet. The outcome assessor is masked because donation-related data is recorded by blood collection staff who are unaware that donors may be participants in a study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fear Control (No Intervention): Participants who report blood donation-related fear who are assigned to this study arm will answer several questions then proceed through the normal blood donation process.
- Fear Intervention (Experimental): Participants who report blood donation-related fear who are assigned to this study arm will answer several questions and view a brief presentation of coping strategies presented via a computer tablet. They will then proceed through the normal blood donation process.
  Interventions: Behavioral: Fear Intervention
- No Fear Control (No Intervention): Participants who report no blood donation-related fear will proceed through the normal blood donation process.

INTERVENTIONS:
Behavioral: Fear Intervention — Coping information related to the fear that was identified by the participant will be presented via a computer tablet.
  Arms: Fear Intervention

SUMMARY:
In this study, high school donors will be asked about their blood donation-related fears prior to their donation. Half of the donors reporting fear will be assigned to a brief coping skills intervention.

DETAILED DESCRIPTION:
In this study the investigators will ask high school donors about their blood donation-related fears prior to their donation. Among those who report donation fear, half will be randomly assigned to receive a brief presentation of coping strategies administered via a computer tablet. The investigators will compare reaction rates and return behavior for the donors and high school drives where the study was conducted to the reaction and retention rates from similar blood drives where no data was collected. The investigators will also examine whether asking about the specific types of fear improves the prediction of syncopal or presyncopal reactions beyond the predictive value of a single fear question. Finally, the investigators will examine whether providing coping information to help manage the fear improves syncopal reaction rates and/or donor retention rates among fearful donors.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for inclusion in this study, the individual must have presented to donate blood at a New York Blood Center high school blood drive where data is being collected and have passed the health screening process.

Exclusion Criteria:

* Less than 16 years of age; inability to read and comprehend English

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4035 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Repeat Blood Donation Attempts | two years post-donation
  Donor records will be used to track subsequent donation attempts during the follow-up.

SECONDARY OUTCOMES:
Blood Donation Confidence | immediately pre-donation
  Confidence in ability to cope with any donation-related fear
Vasovagal Reactions to Blood Donation | immediately post-donation
  phlebotomist ratings of blood donor vasovagal reactions

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R France, PhD, Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No